CLINICAL TRIAL: NCT06526871
Title: Evaluation of Treatment Outcome of Lower Incisors Crowding Using Clear Aligners With Laser Acceleration (Randomized Control Study) .
Brief Title: Evaluation of Treatment Outcome of Lower Incisors Crowding Using Clear Aligners With Laser Acceleration .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huda Abdelhakim (Other Government)
Responsible Party: Sponsor-Investigator, Huda Abdelhakim, Doctor, Faculty of Dental Medicine for Girls
Organization: Faculty of Dental Medicine for Girls (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORTHO-109-2-K
Record Dates: First submitted 2024-07-19; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Tooth Movement
Keywords: Aligner; Crowding; Laser
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control group (Active Comparator): ten patients treated with removable clear aligner
  Interventions: Procedure: clear aligner therapy
- Experimental group (Experimental): ten patients treated with removable clear aligner with application of Low-Level-Laser
  Interventions: Procedure: Low-Level Laser acceleration; Procedure: clear aligner therapy

INTERVENTIONS:
Procedure: Low-Level Laser acceleration — This intervention involves the application of Low-Level Laser Therapy (LLLT) using the Epic X device for patients undergoing orthodontic treatment. The protocol is designed to assess the effects of LLLT on pain reduction and treatment efficacy during the initial leveling and alignment phase of orthodontic therapy using clear aligners .
  Arms: Experimental group
Procedure: clear aligner therapy — Clear aligner therapy involves using a series of custom-made, clear plastic aligners to gradually move teeth into their desired positions. These aligners are worn over the teeth and are typically changed every week as the teeth gradually shift. The treatment process starts with a digital scan or impression of the teeth, which is used to create a 3D model. This model helps in planning the precise movements needed to achieve proper alignment. Throughout the treatment, patients visit their orthodontist periodically to monitor progress and receive new sets of aligners. Clear aligners are popular for their aesthetic appeal and the convenience they offer compared to traditional braces.

SUMMARY:
The present study will be performed to evaluate the effect of low-level laser therapy (LLLT) on the rate of orthodontic tooth movement through the correction of lower incisors crowding using clear aligners

DETAILED DESCRIPTION:
This study will employ a two-arm parallel randomized clinical trial design with an allocation ratio of 1:1. The study will include participants aged 16 to 23 years with mild to moderate anterior lower crowding and Class I Angle malocclusion, presenting with a full set of teeth excluding wisdom teeth. Eligible participants will be randomly assigned to either the intervention group, receiving LLLT in addition to clear aligner therapy, or the control group, receiving clear aligner therapy alone.

Intervention:

The intervention group will undergo LLLT using the Biolase Epic X device, calibrated to 0.2 W power, 0.16 J energy, and 0.8 seconds pulse duration per point. The laser will be applied to five points on the buccal surface (cervical mesial, distal, middle root, apical mesial, and distal) and four points on the lingual surface (cervical mesial, distal, middle root, and middle apical) of the target tooth. LLLT sessions will be conducted weekly over seven sessions.

ELIGIBILITY:
Inclusion Criteria:

1. A well-behaved, compliant, and motivated patient.
2. Patients from 16 to 23 years old .
3. Patients with mild to moderate anterior lower crowding.
4. Full complement of teeth (except for wisdom teeth).
5. Class I Angle malocclusion .

Exclusion Criteria:

1. Patients with missed anterior teeth .
2. Class II or III Malocclusion (dental or skeletal ) .
3. Any systemic diseases that may interfere with assigned treatment plan .
4. Periodontal affection especially at lower anterior teeth .

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
• Little irregularity index | through study completion, an average of 6 months
  The Little Irregularity Index is a quantitative method used to assess the degree of dental crowding. It measures the linear displacement of the contact points of the mandibular anterior teeth (canine to canine) from their ideal positions. This measurement is taken before and after orthodontic treatment using scanned 3D models, allowing for an objective evaluation of alignment improvement.

SECONDARY OUTCOMES:
• Treatment time | through study completion, an average of 6 months
  The duration of orthodontic treatment, including active treatment phases such as wearing aligners or undergoing procedures like interproximal reduction, is crucially monitored. This active treatment time is distinct from overall treatment duration, which encompasses intervals such as retention phases or breaks between aligner changes.
• Number of aligners | through study completion, an average of 6 months
  The number of aligners measurement involves determining the total quantity of clear aligners required for a patient's orthodontic treatment.
• Patient comfort and satisfaction | through study completion, an average of 6 months
  Patient comfort and satisfaction were evaluated using standardized scales, including Visual Analog Scales (VAS) , to assess pain levels, oral discomfort, and overall treatment experience.
• Refinement rate | through study completion, an average of 6 months
  The refinement rate in orthodontics refers to the frequency and extent of adjustments made to aligners or appliances during treatment to achieve optimal tooth alignment. It is typically measured by assessing the need for additional aligners,
• Digital cast accuracy | through study completion, an average of 6 months
  Digital cast accuracy was assessed using 3D surface comparison methods, comparing intraoral scans with traditional plaster models.
• Tooth movement accuracy | through study completion, an average of 6 months
  This process involved aligning and overlaying 3D models to assess the extent and direction of tooth displacement over time.
• Software predictability | through study completion, an average of 6 months
  3D models were superimposed to analyze the accuracy of predicted tooth movements compared to actual outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Samir A Ibrahim, professor, Principal Investigator — Al-Azhar University
Locations (1):
- AL-Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Das PJ, Dkhar W, Pradhan A. An Evaluation of Dental Crowding in Relation to the Mesiodistal Crown Widths and Arch Dimensions in Southern Indian Population. J Clin Diagn Res. 2017 Sep;11(9):TC10-TC13. doi: 10.7860/JCDR/2017/29642.10554. Epub 2017 Sep 1. PMID 29207804
- [Background] Jaber ST, Hajeer MY, Burhan AS, Latifeh Y. The Effect of Treatment With Clear Aligners Versus Fixed Appliances on Oral Health-Related Quality of Life in Patients With Severe Crowding: A One-Year Follow-Up Randomized Controlled Clinical Trial. Cureus. 2022 May 30;14(5):e25472. doi: 10.7759/cureus.25472. eCollection 2022 May. PMID 35663697
- [Background] Knosel M, Nuser C, Jung K, Helms HJ, Engelke W, Sandoval P. Interaction between deglutition, tongue posture, and malocclusion: A comparison of intraoral compartment formation in subjects with neutral occlusion or different types of malocclusion. Angle Orthod. 2016 Sep;86(5):697-705. doi: 10.2319/101615-699.1. Epub 2016 Feb 19. PMID 26894981
- [Background] Tamer I, Oztas E, Marsan G. Orthodontic Treatment with Clear Aligners and The Scientific Reality Behind Their Marketing: A Literature Review. Turk J Orthod. 2019 Dec 1;32(4):241-246. doi: 10.5152/TurkJOrthod.2019.18083. eCollection 2019 Dec. PMID 32110470
- [Background] Hennessy J, Garvey T, Al-Awadhi EA. A randomized clinical trial comparing mandibular incisor proclination produced by fixed labial appliances and clear aligners. Angle Orthod. 2016 Sep;86(5):706-12. doi: 10.2319/101415-686.1. PMID 27571371
- [Background] Baghizadeh Fini M, Olyaee P, Homayouni A. The Effect of Low-Level Laser Therapy on the Acceleration of Orthodontic Tooth Movement. J Lasers Med Sci. 2020 Spring;11(2):204-211. doi: 10.34172/jlms.2020.34. Epub 2020 Mar 15. PMID 32273964
- [Background] Sharma R, Drummond R, Wiltshire W, Schroth R, Lekic M, Bertone M, Tate R. Quality of life in an adolescent orthodontic population. Angle Orthod. 2021 Nov 1;91(6):718-724. doi: 10.2319/062820-592.1. PMID 34260709
- [Background] Ghaffar YKA, El Sharaby FA, Negm IM. Effect of low-level laser therapy on the time needed for leveling and alignment of mandibular anterior crowding. Angle Orthod. 2022 Jul 1;92(4):478-486. doi: 10.2319/102721-795.1. PMID 35344012
- [Background] Soares Bonato RC, Abel Mapengo MA, de Azevedo-Silva LJ, Janson G, de Carvalho Sales-Peres SH. Tooth movement, orofacial pain, and leptin, interleukin-1beta, and tumor necrosis factor-alpha levels in obese adolescents. Angle Orthod. 2022 Jan 1;92(1):95-100. doi: 10.2319/011321-44.1. PMID 34338736
- [Background] Bakdach WMM, Hadad R. Effectiveness of low-level laser therapy in accelerating the orthodontic tooth movement: A systematic review and meta-analysis. Dent Med Probl. 2020 Jan-Mar;57(1):73-94. doi: 10.17219/dmp/112446. PMID 32314880
- [Background] Cossetin E, Janson G, de Carvalho MG, de Carvalho RA, Henriques JF, Garib D. Influence of low-level laser on bone remodeling during induced tooth movement in rats. Angle Orthod. 2013 Nov;83(6):1015-21. doi: 10.2319/100812-789.1. Epub 2013 May 14. PMID 23672280
- [Background] Guram G, Reddy RK, Dharamsi AM, Syed Ismail PM, Mishra S, Prakashkumar MD. Evaluation of Low-Level Laser Therapy on Orthodontic Tooth Movement: A Randomized Control Study. Contemp Clin Dent. 2018 Jan-Mar;9(1):105-109. doi: 10.4103/ccd.ccd_864_17. PMID 29599594
- [Background] 13. Cokakoglu S. , Aydoğan F. Aydın B. low level laser therapy in orthodontics . Meandros Med Dent J.2018;19:99-105 .
- [Background] AlSayed Hasan MMA, Sultan K, Hamadah O. Low-level laser therapy effectiveness in accelerating orthodontic tooth movement: A randomized controlled clinical trial. Angle Orthod. 2017 Jul;87(4):499-504. doi: 10.2319/062716-503.1. Epub 2016 Nov 21. PMID 27869476
- [Background] 15. Ponciano F. A. S. , Gutiérrez-Rojo M. F. , Gutiérrez-Rojo J. F. .Crowding severity associated with dental mass . Revista Mexicana de Ortodoncia .2016;4:165-8 .
- [Background] Masucci C, Oueiss A, Maniere-Ezvan A, Orthlieb JD, Casazza E. [What is a malocclusion?]. Orthod Fr. 2020 Jun 1;91(1-2):57-67. doi: 10.1684/orthodfr.2020.11. French. PMID 33146134

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT06526871/Prot_SAP_000.pdf